CLINICAL TRIAL: NCT00950898
Title: Human Trial of the Acute Effects of Coffee on Glucose Metabolism
Brief Title: The Acute Effects of Coffee on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooklyn College of the City University of New York (Other)
Responsible Party: James Greenberg, PhD., Principal Investigator, Brooklyn College of the City University of New York
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 07-020
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
Keywords: coffee; caffeine; glucose metabolism; insulin sensitivity; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: decaff — 2 mugs of decaffeinated coffee
Other: caffcoff — 2 mugs of caffeinated coffee
Other: caffeine — 2 mugs of hot water containing caffeine
Other: placebo — 2 mugs of hot water

SUMMARY:
The purpose of this study was to determine the acute effects of decaffeinated coffee, caffeinated coffee and caffeine on glucose metabolism in humans

ELIGIBILITY:
Inclusion Criteria:

* healthy young males
* nonsmokers
* moderate alcohol users

Exclusion Criteria:

* not on any medications that could alter glucose metabolism
* no history of blood disorders

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
plasma glucose levels | 0, 10, 30, 60, 90, and 120 minutes.

SECONDARY OUTCOMES:
plasma insulin | 0, 10, 30, 60, 90, and 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: James Greenberg, Ph.D., Principal Investigator — Brooklyn College of the City University of New York
Locations (1):
- Brooklyn College of the City University of New York, Brooklyn, New York, United States